CLINICAL TRIAL: NCT00001497
Title: Assessment of Attentional Functioning in Children With HIV-1 Infection
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960030; 96-C-0030
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity; HIV Infections; Paralysis
Keywords: Brain Imaging; Encephalopathy; Hyperactivity; Neuroimmunology; Reaction Time Tasks
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; HIV Infections; Paralysis; Brain Diseases; Spasm

SUMMARY:
Children with symptomatic HIV-1 (Human Immunodeficiency Virus) infection are at increased risk for developing severely disabling neurological and neuropsychological deficits. HIV-1 related CNS (Central Nervous System) disease is a clinical syndrome, manifested by varying and sometimes discordant degrees of cognitive, motor and behavioral impairment. A continuum of clinical presentations attributed to the effects of HIV-1 infection on the CNS, ranging from apparently normal development, decreases in the rate of new learning to the loss of acquired skills have been observed. Two domains of psychological functioning appear most susceptible to the effects of HIV infection on the central nervous system in children: expressive behavior and attentional processes (Brouwers, et al, 1994).

Attention deficits have been documented as a relative weakness on the "freedom from distractibility" subclass of IQ tests (Brouwers et al, 1989) and on behavior assessment (Moss et al, 1994). Attention, however, has many subcomponents such as focused attention, divided attention, vigilance, etc. Direct assessment of attentional functioning using reaction time has not yet been conducted and questions whether attentional components are differentially affected by the virus have not been addressed.

The proposed study would assess different components of attentional functioning in children with HIV-1 disease. A quantitative and systematic method is developed that could complement the existing standardized instruments used for measuring attention and neurocognitive function in this population. Simple alerted visual reaction time will be measured with varying preparatory intervals, a two-choice reaction time in a go/no-go paradigm will be administered, and a continuous performance, divided reaction time test and an object decision task will be given. Performance on these measures will also be related to measures of brain structure and stage of HIV-1 disease.

DETAILED DESCRIPTION:
Children with symptomatic HIV-1 (Human Immunodeficiency Virus) infection are at increased risk for developing severely disabling neurological and neuropsychological deficits. HIV-1 related CNS (Central Nervous System) disease is a clinical syndrome, manifested by varying and sometimes discordant degrees of cognitive, motor and behavioral impairment. A continuum of clinical presentations attributed to the effects of HIV-1 infection on the CNS, ranging from apparently normal development, decreases in the rate of new learning to the loss of acquired skills have been observed. Two domains of psychological functioning appear most susceptible to the effects of HIV infection on the central nervous system in children: expressive behavior and attentional processes (Brouwers, et al, 1994).

Attention deficits have been documented as a relative weakness on the "freedom from distractibility" subclass of IQ tests (Brouwers et al, 1989) and on behavior assessment (Moss et al, 1994). Attention, however, has many subcomponents such as focused attention, divided attention, vigilance, etc. Direct assessment of attentional functioning using reaction time has not yet been conducted and questions whether attentional components are differentially affected by the virus have not been addressed.

The proposed study would assess different components of attentional functioning in children with HIV-1 disease. A quantitative and systematic method is developed that could complement the existing standardized instruments used for measuring attention and neurocognitive function in this population. Simple alerted visual reaction time will be measured with varying preparatory intervals, a two-choice reaction time in a go/no-go paradigm will be administered, and a continuous performance, divided reaction time test and an object decision task will be given. Performance on these measures will also be related to measures of brain structure and stage of HIV-1 disease.

ELIGIBILITY:
Children and adolescents with HIV infection ages 5-18.

Have to be on another treatment protocol at the Division of Clinical Sciences, NCI.

No children with non-HIV associated CNS compromise, such as for example resulting from head trauma, or genetic factors.

No children with uncorrectable (20/20) vision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1995-12; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Brouwers P, Riccardi R, Poplack D, Fedio P. Attentional deficits in long-term survivors of childhood acute lymphoblastic leukemia (ALL). J Clin Neuropsychol. 1984 Aug;6(3):325-36. doi: 10.1080/01688638408401222. PMID 6590573
- [Background] Brouwers P, DeCarli C, Civitello L, Moss H, Wolters P, Pizzo P. Correlation between computed tomographic brain scan abnormalities and neuropsychological function in children with symptomatic human immunodeficiency virus disease. Arch Neurol. 1995 Jan;52(1):39-44. doi: 10.1001/archneur.1995.00540250043011. PMID 7826274
- [Background] DeCarli C, Civitello LA, Brouwers P, Pizzo PA. The prevalence of computed tomographic abnormalities of the cerebrum in 100 consecutive children symptomatic with the human immune deficiency virus. Ann Neurol. 1993 Aug;34(2):198-205. doi: 10.1002/ana.410340216. PMID 8338344